CLINICAL TRIAL: NCT03392779
Title: A Phase 1 Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ZSP1601 and the Effect of Food on ZSP1601 Pharmacokinetics in Chinese Healthy Subjects.
Brief Title: Study in Chinese Healthy Adults to Evaluate the Safety, Tolerability and Pharmacokinetics on ZSP1601, and the Effect of Food on ZSP1601 Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Zhongsheng Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZSP1601-16-01
Record Dates: First submitted 2018-01-02; First posted 2018-01-08 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking for Participant, Investigator and Clinical Research Associate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- ZSP1601(single dose)-25 mg while fasted(Cohort 1) (Experimental): ZSP1601 25 mg /Placebo
  Interventions: Drug: ZSP1601 25 mg; Drug: Placebo 25mg
- ZSP1601(single dose)-50 mg while fasted(Cohort 2) (Experimental): ZSP1601 50 mg/Placebo
  Enrollment into Cohort 2 will begin upon assurance of safety for Cohort 1.
  Interventions: Drug: ZSP1601 50 mg; Drug: Placebo 50 mg
- ZSP1601(single dose)-100 mg while fasted(Cohort 3) (Experimental): ZSP1601 100 mg/Placebo
  Enrollment into Cohort 3 will begin upon assurance of safety for Cohort 2.
  Interventions: Drug: ZSP1601 100 mg; Drug: Placebo 100 mg
- ZSP1601(single dose)-175 mg while fasted(Cohort 4) (Experimental): ZSP1601 175 mg/Placebo
  Enrollment into Cohort 4 will begin upon assurance of safety for Cohort 3.
  Interventions: Drug: ZSP1601 175 mg; Drug: Placebo 175 mg
- ZSP1601(single dose)-275 mg while fasted(Cohort 5,i.e.Group A) (Experimental): ZSP1601 275 mg/Placebo
  Enrollment into Cohort 5 will begin upon assurance of safety for Cohort 4.
  Interventions: Drug: ZSP1601 275 mg; Drug: Placebo 275 mg
- ZSP1601(single dose)-350 mg while fasted(Cohort 6) (Experimental): ZSP1601 350 mg/Placebo
  Enrollment into Cohort 6 will begin upon assurance of safety for Cohort 5.
  Interventions: Drug: ZSP1601 350 mg; Drug: Placebo 350mg
- ZSP1601(food effect)-100 mg (Cohort FE) (Experimental): Period 1 (Day1 to Day4): Group A and Group B receive ZSP1601 100 mg/Placebo under the fasting or fed condition ,respectively on Day1.
  Period 2 (Day 8 to Day11): Group A and Group B receive ZSP1601 100 mg/Placebo under the fed or fasting condition ,respectively on Day8.
  Interventions: Drug: ZSP1601 100 mg; Drug: Placebo 100mg
- ZSP1601(multiple doses)-50 mg (Cohort 7) (Experimental): 50 mg ZSP1601 will be administrated while fasted or fed according to the results of Cohort FE
  ZSP1601 50 mg/Placebo for 14 Days.
  Interventions: Drug: ZSP1601 50 mg; Drug: Placebo 50 mg
- ZSP1601(multiple doses)-100 mg (Cohort 8) (Experimental): Enrollment into Cohort 8 will begin upon assurance of safety for Cohort 7.
  ZSP1601 100 mg/Placebo for 14 Days.
  Interventions: Drug: ZSP1601 100 mg; Drug: Placebo 100 mg

INTERVENTIONS:
Drug: ZSP1601 25 mg — ZSP1601 tablet administered orally once daily under fasted condition
  Arms: ZSP1601(single dose)-25 mg while fasted(Cohort 1)
Drug: Placebo 25mg — Participants will receive placebo matching to ZSP1601 orally once daily under fasted condition
  Arms: ZSP1601(single dose)-25 mg while fasted(Cohort 1)
Drug: ZSP1601 50 mg — ZSP1601 tablet administered orally once daily under fasted condition
  Arms: ZSP1601(single dose)-50 mg while fasted(Cohort 2)
Drug: Placebo 50 mg — Participants will receive placebo matching to ZSP1601 orally once daily under fasted condition
  Arms: ZSP1601(single dose)-50 mg while fasted(Cohort 2)
Drug: ZSP1601 100 mg — ZSP1601 tablets administered orally once daily in the fasting state
  Arms: ZSP1601(single dose)-100 mg while fasted(Cohort 3)
Drug: Placebo 100 mg — Participants will receive placebo matching to ZSP1601 orally once daily in the fasting state
  Arms: ZSP1601(single dose)-100 mg while fasted(Cohort 3)
Drug: ZSP1601 175 mg — ZSP1601 tablets administerekd orally once daily under fasted condition
  Arms: ZSP1601(single dose)-175 mg while fasted(Cohort 4)
Drug: Placebo 175 mg — Participants will receive placebo matching to ZSP1601 orally once daily under fasted condition
  Arms: ZSP1601(single dose)-175 mg while fasted(Cohort 4)
Drug: ZSP1601 275 mg — ZSP1601 tablets administered orally once daily in the fasting state
  Arms: ZSP1601(single dose)-275 mg while fasted(Cohort 5,i.e.Group A)
Drug: Placebo 275 mg — Participants will receive placebo matching to ZSP1601 orally once daily in the fasting state
  Arms: ZSP1601(single dose)-275 mg while fasted(Cohort 5,i.e.Group A)
Drug: ZSP1601 350 mg — ZSP1601 tablets administered orally once daily under fasted condition
  Arms: ZSP1601(single dose)-350 mg while fasted(Cohort 6)
Drug: Placebo 350mg — Participants will receive placebo matching to ZSP1601 orally once daily under fasted condition
  Arms: ZSP1601(single dose)-350 mg while fasted(Cohort 6)
Drug: ZSP1601 100 mg — ZSP1601 tablets administered orally once daily under fasted or fed condition
  Arms: ZSP1601(food effect)-100 mg (Cohort FE)
Drug: Placebo 100mg — Participants will receive placebo matching to ZSP1601 orally once daily under fasted or fed condition
  Arms: ZSP1601(food effect)-100 mg (Cohort FE)
Drug: ZSP1601 50 mg — ZSP1601 tablets administered orally once daily under fasted or fed condition due to the results of Cohort FE for 14 Days(a total of 14 doses).
  Arms: ZSP1601(multiple doses)-50 mg (Cohort 7)
Drug: Placebo 50 mg — Participants will receive placebo matching to ZSP1601 orally once daily under fasted or fed condition due to the results of Cohort FE for 14 Days(a total of 14 doses).
  Arms: ZSP1601(multiple doses)-50 mg (Cohort 7)
Drug: ZSP1601 100 mg — ZSP1601 tablets administered orally once daily under fasted or fed condition due to the results of Cohort FE for 14 Days(a total of 14 doses).
  Arms: ZSP1601(multiple doses)-100 mg (Cohort 8)
Drug: Placebo 100 mg — Participants will receive placebo matching to ZSP1601 orally once daily under fasted or fed condition due to the results of Cohort FE for 14 Days(a total of 14 doses).
  Arms: ZSP1601(multiple doses)-100 mg (Cohort 8)

SUMMARY:
This study will evaluate the safety, tolerability and pharmacokinetics (PK) of escalating single- and multiple-oral doses of ZSP1601 on fasted condition, and characterize PK of ZSP1601 on an empty stomach (fasted condition) and following a high fat, high calorie meal (fed condition) in a 2-period, 2-sequence manner. The study will be conducted in 3 parts (Ascending single dose, multiple dose and food effect). Participants will receive either ZSP1601 or placebo .

DETAILED DESCRIPTION:
The study is a randomized, double-blind phase 1 trial including 3 parts: single ascending dose(SAD) part,multiple ascending dose(MAD) part and postprandial pharmacokinetics part.The primary aims of the study as below:

Evaluating the safety and tolerance of single and multiple dose of ZSP1601 in healthy volunteers.

Evaluating the fasting and postprandial pharmacokinetic parameters of ZSP1601 in healthy volunteers.

Eligible participants will be admitted to the trial center on Day -1. Subjects will be randomly assigned to either experimental groups or placebo groups, according to a randomisation schedule in a (4:1) ratio (8 in per experimental group). Subjects in SAD will receive 25、50、100、175、275、350 mg once daily respectively.Each dose will be administrated after assurance of safety for the former dose. Subjects in MAD will receive 50 or 100 mg once daily for 14days respectively.The treatment in food effect consists of 2 periods,and subjects will receive 100mg on fasting and postprandial states respectively. There will be a 7-day wash out period between treatment periods.To monitor AEs,record abnormalities (12-lead ECG,Vital signs,Physical examination,Clinical Laboratory),and detect the pharmacokinetics of ZSP1601.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are required to meet the following criteria in order to be included in the trial:

  1. Signature of a dated Informed Consent Form (ICF) indicating that the subject has been informed of all the relevant aspects(including adverse events) of the trial prior to enrollment.
  2. Subjects must be willing and able to adhere to the visit schedule and protocol requirements and be available to complete the study.
  3. Subjects(including partners)have no gestation plans and must use reliable methods of contraception during the study and until 6 months following the last dose of investigational product.
  4. Males and female subjects between 18-50 years (Both inclusive).
  5. Body weight is no less than 50kg in males and no less than 45kg in females.Body mass index (BMI) 18≤BMI≤28 kg/m2; BMI is determined by the following equation: BMI = weight/height2 (kg/m2).
  6. Physical condition:No significant abnormalities in medical history, including cardiovascular system, liver, kidneys, gastrointestinal system, neural system, respiratory system (eg.asthma,asthma induced by exercise,chronic obstructive pulmonary disease), mental, metabolism, etc.
  7. Subjects in general good health or No significant abnormalities in the opinion of the investigator as determined by vital signs and a physical examination.

Exclusion Criteria:

* Eligible subjects must not meet any of the following exclusion criteria:

  1. The average daily smoking are more than 5 cigarettes within 3 months prior to screening.
  2. Known hypersensitivity and/or allergy to some drugs and food.
  3. Known history of drug or alcohol abuse.(defined as consumption of 14 units of alcohol per week:1 unit=285ml of beer; or the equivalent of 25ml of spirit, or 100ml of wine )
  4. Subjects who donated blood or bleeding profusely(> 400 mL)in the 3 months preceding study screening.
  5. Dysphagia or any medical history in gastrointestinal that interferes with the absorption of drugs.
  6. History or presence of any disease or condition known to increase the risk of bleeding, eg.acute gastritis, duodenal ulcer, etc.
  7. Frequently suffers from postural hypotension.
  8. History of frequent nausea or vomit causes by any etiology.
  9. Concomitant therapy with any drugs with known hepatic enzyme-inducing or inhibiting agents that may change the activity of CYP3A4 prior to screening or during the study.
  10. Use of any prescription or over-the-counter (OTC) medications, vitamins and herbal or dietary supplements within 14 days prior to screening.
  11. History of having any special food(including dragon fruit,mango,grapefruit,etc.),strenuous exercises,or other factors may interfere with the absorption, distribution, metabolism, or excretion of drug within 14 days prior to screening.
  12. Subjects with recent significant change in diet or exercise .
  13. Participated in another clinical research study and received any investigational products within 3 months prior to dosing.
  14. Inability to consume the food provided in the study ( a high fat, high calorie meal includes two eggs for 100g, bacon 20g, a butter toast for 50g, french fries for 115g, whole milk for 240ml).This requirement only applies to subjects under fed condition.
  15. Presence of clinically significant abnormalities in ECG or QTc>470ms in males,or QTc>480ms in females.
  16. Pregnancy or breastfeeding at screening and during the study.All female subjects of childbearing potential must have a negative urine pregnancy test at screening and during the trial.
  17. Any clinically significant abnormality upon physical examination or in the clinical laboratory tests. History or presence of a clinically significant gastrointestinal, renal, hepatic, neurologic, hematic, endocrine, neoplastic, pulmonary, immune, psychiatric or cardiovascular and cerebrovascular disorder(s) (but not limited to above disorders).
  18. Presence of human immunodeficiency virus (HIV), viral hepatitis(including hepatitis C virus (HCV) or hepatitis B virus (HBV) ),treponema pallidum antibodies at screening.
  19. Any acute illness or concomitant medication from screening to first dosing.
  20. Have chocolate, any food or beverage that contains caffeine or xanthine within 24 hours prior to dosing.
  21. Take any product contains alcohol within 24 hours prior to dosing.
  22. Positive for urine drug screening or history of substance abuse for a period of 5 consecutive years before screening.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Number and severity of treatment-emergent adverse events (TEAEs) and Serious Adverse Events(SAE) following oral doses(single,multiple and food effect)of ZSP1601 and placebo. | SAD Group: Up to 4 days, MAD: Up to 17days, FE group: Up to 11 days after first dose
Concomitant Medication | UP to 4, 17, 11 days for SAD, MAD, FE part respectively
Clinical Laboratory Abnormalities(Blood routine test, serum biochemical test, conventional coagulation examinations, urine examination ) post dose of ZSP1601 and placebo. | UP to 4, 17, 11 days for SAD, MAD, FE part respectively
12-lead ECG Abnormalities following oral dosing of ZSP1601 and placebo. | UP to 4, 17, 11 days for SAD, MAD, FE part respectively
Vital signs Abnormalities following oral dosing of ZSP1601 and placebo. | UP to 4, 17, 11 days for SAD, MAD, FE part respectively
Physical examination Abnormalities following oral dossing of ZSP1601 and placebo. | UP to 4, 17, 11 days for SAD, MAD, FE part respectively
Cardiac color ultrasound(UCG) Abnormalities following multiple oral doses of ZSP1601 and placebo. | Screening, Day17

SECONDARY OUTCOMES:
AUClast（AUC0-t）of ZSP1601 | UP to 2, 16, 9 days for SAD, MAD, FE part respectively
  AUClast is defined as the concentration of drug from time zero to the last quantifiable concentration.
AUCinf（AUC0-∞）of ZSP1601 | UP to 2, 16, 9 days for SAD, MAD, FE part respectively
  AUCinf is defined as the concentration of drug extrapolated to infinite time (area under the plasma concentration versus time curve extrapolated to infinite time).
Cmax of ZSP1601 | UP to 2, 16, 9 days for SAD, MAD, FE part respectively
  Cmax is defined as the maximum observed concentration of drug in plasma.
Tmax of ZSP1601 | UP to 2, 16, 9 days for SAD, MAD, FE part respectively
  Tmax is defined as the time to maximum concentration.
t1/2z of ZSP1601 | UP to 2, 16, 9 days for SAD, MAD, FE part respectively
  t1/2z is defined as the time to decline half of the drug concentration in plasma.
Single-dose PK Parameter: Ae of ZSP1601 | Up to Day 2 post-dose
  Ae is defined as the amount of unchanged drug excreted in urine or faeces after administration.
Single-dose PK Parameter: Fe0-t of ZSP1601 | Up to Day 2 post-dose
  Fe0-t is defined as the cumulative excretion rate of the drug in urine and feces.
CL/F of ZSP1601 | UP to 2, 16, 9 days for SAD, MAD, FE part respectively
  CL/F is defined as the ratio of total clearance(Cl) to bioavailability(F).
λz of ZSP1601 | UP to 2, 16, 9 days for SAD, MAD, FE part respectively
  λz is defined as the ratio between the elimination of compound per unit time and the total amount of compound.
CLr of ZSP1601 | UP to 2, 16, 9 days for SAD, MAD, FE part respectively
  CLr is defined as how many milliliters of plasma in which some substance can be completely eliminated in the unit time (per minute) of two kidneys
Multiple-dose plasma PK parameter: Rac of ZSP1601 at steady state | Up to 16days
  Rac (Accumulation Index) is defined as the ratio between AUC0-XX in Day XX and AUC0-XX in Day1
Multiple-dose plasma PK parameter: DF of ZSP1601 at steady state | Up to 16 days
  DF is defined as the percentage of fluctuation in steady state is 100 * (Cmax, ss - Cmin, ss)/Cavg, ss.
Multiple-dose plasma PK parameter: Cmin of ZSP1601 at steady state | Up to 16days
  Cmin is defined as the minimum observed concentration of drug in plasma at steady state.

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, MD, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Derived] Zhu X, Wu M, Wang H, Li H, Lin J, Peng Y, Hu Y, Li C, Ding Y. Safety, tolerability, and pharmacokinetics of the novel pan-phosphodiesterase inhibitor ZSP1601 in healthy subjects: a double-blinded, placebo-controlled first-in-human single-dose and multiple-dose escalation and food effect study. Expert Opin Investig Drugs. 2021 May;30(5):579-589. doi: 10.1080/13543784.2021.1900822. Epub 2021 Mar 25. PMID 33682556